CLINICAL TRIAL: NCT00737126
Title: Folic Acid Administration Reduces the Progression of Microalbuminuria
Brief Title: The Effect of Folic Acid Administration in the Progression of Microalbuminuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Laboratorios Valdecasas S.A. (Unknown)
Responsible Party: Jesús Zacarías Villarreal Pérez, Departamento de Endocrinologia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endo02
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Diabetic Nephropathies; Hyperhomocysteinemia
Keywords: Diabetic nephropathies; Hyperhomocysteinemia; Folic acid; Endothelial dysfunction
MeSH Terms: conditions — Diabetic Nephropathies; Hyperhomocysteinemia | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Administration of an oral placebo pill
  Interventions: Drug: Placebo
- 2 (Experimental): Administration of oral folic acid
  Interventions: Drug: Folic acid

INTERVENTIONS:
Drug: Folic acid — Administration of a daily tablet containing 5 mg of folic acid for 4 months.
  Arms: 2
Drug: Placebo — Administration of an oral placebo pill
  Arms: 1

SUMMARY:
The development of diabetic nephropathy has been linked to several genetic polymorphisms, including those related with homocysteine metabolism such as the methylenetetrahydrofolate reductase (MTHFR)and the cystathionine-beta-synthase genes. Such alterations are associated with hyperhomocysteinemia, which is a known independent risk factor for the development of endothelial dysfunction and cardiovascular disease.

In the Mexican population there is a high prevalence of the C677T MTHFR mutation. The investigators performed this study to evaluate the prevalence of this polymorphism in type 2 diabetic patients with diabetic nephropathy compared with type 2 diabetic patients without nephropathy, besides evaluating the relationship of hyperhomocysteinemia with endothelial dysfunction and microalbuminuria before and after the administration of folic acid. We proposed that the endothelial dysfunction caused by the hyperhomocysteinemia could be reversed after the administration of folic acid.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients with 5 to 15 years of diagnosis
* Microalbuminuria (defined as a urinary albumin/creatinine ratio between 30 and 300 mg/g)
* A1c less than 9% in the last year

Exclusion Criteria:

* Acute diabetic complications
* A1c greater than 9% in the last year
* Acute infectious process
* Hepatic disease
* Thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in albumin excretion rate | Four months

SECONDARY OUTCOMES:
Change in serum homocysteine, thrombomodulin and von Willebrand factor. | Four months.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Lavalle, MD, Study Chair — Departamento de Endocrinología del Hospital Universitario "José E. González"
Locations (1):
- Hospital Universitario "José E. González", Monterrey, Nuevo León, Mexico